CLINICAL TRIAL: NCT02498795
Title: Comparative Research Among 3 Action Protocol in Other to Approach Chronic Patellar Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Universidad San Jorge (Other)
Responsible Party: Principal Investigator, Maria Pilar López Royo, Graduate, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P115/0017
Record Dates: First submitted 2015-06-06; First posted 2015-07-15 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Tendinopathy
Keywords: Intratissue Percutaneous Electrolysis; Dry needling; Eccentric exercise; Patella
MeSH Terms: conditions — Tendinopathy; Patella Fracture | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group of Dry Needling (Active Comparator): They will receive a treatment of dry needling with ultrasound scan together with a treatment in which they will realize eccentric exercise's program that the patient will have to realize in his domicile.
  The needle will get in the relevant zone of treatment. The punction will be realized using the technique of entry - Hong's rapid exit. Three punction will realize in the disabled zone of 3 seconds of duration.
  Interventions: Other: Group of Dry Needling
- Group of electrolysis (Active Comparator): They will receive a treatment of Intratissue Percutaneous Electrolysis with ultrasound scan together with a treatment in which they will realize eccentric exercise's program that the patient will have to realize in his domicile.
  The needle will get in the relevant zone of treatment. An intensity of 3 milliampere will be in use, during 3 seconds and one will repeat 3 times.
  Interventions: Other: Group of Electrolysis
- Control Group (Placebo Comparator): They will receive a treatment of punction placebo with ultrasound scan together with a treatment in the one that will realize eccentric exercise's program that the patient will have to realize in his domicile.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Group of Dry Needling — Every group will receive a total of 4 treatment distributed throughout 8 weeks of treatment. The program of eccentric exercises that will have to realize it in his domicile every day.
  Arms: Group of Dry Needling
Other: Group of Electrolysis — Every group will receive a total of 4 treatment distributed throughout 8 weeks of treatment. The program of eccentric exercises that will have to realize it in his domicile every day.
  Arms: Group of electrolysis
Other: Control Group — Every group will receive a total of 4 treatment distributed throughout 8 weeks of treatment. The program of eccentric exercises that will have to realize it in his domicile every day.
  Arms: Control Group

SUMMARY:
The accomplishment of a treatment with Intratissue Percutaneous Electrolysis of additional form to the accomplishment of eccentric exercise's program in patients with chronic patellar tendinopathy is more effective than the accomplishment of an additional treatment with dry needling or eccentric exercise's program realized of isolated form.

DETAILED DESCRIPTION:
Experimental study randomized with double blind, whose purpose is to compare three protocols in those who apply different protocols of physical therapy to themselves in three groups of intervention with patients with chronic patellar tendinopathy.

There take part in this study young women of both sexes, of Zaragoza and of different sports clubs of entity 18 and 40 years, that they realize of habitual form (minimum 3 times a week) a sport. All of them present chronic patellar tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age understood between 18 and 40 years.
* To practise any sport of habitual form.
* Patients diagnosed of chronic patellar tendinopathy with a minimum of 3 months of evolution and with stable symptomatology.
* Pain to the palpation of the tendon in the low pole of the knee and during the training or competition.
* Punctuation of the questionnaire VISA-P under 80.

Exclusion Criteria:

* Patient had an operation on the knee affected in the last 6 months.
* Infiltrations in the knee affected in the last 3 months.
* Patient who has received pharmacological treatment or physical therapy in the last 48 hours.
* Pathology with less than 3 months of evolution.
* To present bilateral chronic tendinopathy.
* Punctuation of the questionnaire major or equal Visa - p of 80.
* Inability to apply someone of the techniques of treatment or valuation for absolute or relative contraindication.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in functionality at 8 weeks as measured by Visa-p | 8 weeks
  This scale consists of eight questions, the first six questions of which employ an analogical visual scale in order to assign a score of 0 to 10, where 10 represents the optimum state, for the purpose of quantifying pain and function in different activities, whereas the last two questions assess the level of functionality and ability to perform physical activity.

SECONDARY OUTCOMES:
Pain, as measured by Visual Analog Scale | 0, 8 and 20 weeks
  Participants will be explained that a score of 0 indicates the absence of pain whereas a score of 10 represents the maximum tolerable pain
Quality of life by SF-36 | 0, 8 and 20 weeks
  Health Survey
Thickness of the tendon, as measured by ultrasound scan | 0, 8 and 20 weeks
  Tendon structure
Height of the jump | 0, 8 and 20 weeks
  Jump test with a force platform
Concentric force of the low members | 0, 8 and 20 weeks
  Jump test with a force platform
Speed of the jump | 0, 8 and 20 weeks
  Jump test with a force platform
Hypervascularity, as measured by ultrasound scan | 0, 8 and 20 weeks
  Tendon structure
Functionality, as measured by Visa-p | 0 and 20 weeks
  This scale consists of eight questions, the first six questions of which employ an analogical visual scale in order to assign a score of 0 to 10, where 10 represents the optimum state, for the purpose of quantifying pain and function in different activities, whereas the last two questions assess the level of functionality and ability to perform physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Gómez-Trullén, PhD, Study Director — Universidad de Zaragoza; Pablo Herrero, PhD, Study Director — Universidad San Jorge
Locations (1):
- Universidad San Jorge, Villanueva de Gállego, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lopez-Royo MP, Rios-Diaz J, Galan-Diaz RM, Herrero P, Gomez-Trullen EM. A Comparative Study of Treatment Interventions for Patellar Tendinopathy: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 May;102(5):967-975. doi: 10.1016/j.apmr.2021.01.073. Epub 2021 Feb 6. PMID 33556350
- [Derived] Lopez-Royo MP, Gomez-Trullen EM, Ortiz-Lucas M, Galan-Diaz RM, Bataller-Cervero AV, Al-Boloushi Z, Hamam-Alcober Y, Herrero P. Comparative study of treatment interventions for patellar tendinopathy: a protocol for a randomised controlled trial. BMJ Open. 2020 Feb 16;10(2):e034304. doi: 10.1136/bmjopen-2019-034304. PMID 32066608